CLINICAL TRIAL: NCT01973049
Title: A Phase 3 Evaluation of a Daclatasvir/Asunaprevir/BMS-791325 Fixed Dose Combination in Subjects With Genotype 1 Chronic Hepatitis C and Compensated Cirrhosis
Brief Title: UNITY 2: A Study of an Investigational Treatment Regimen of DCV+ASV+BMS-791325 in a Fixed Dose Combination (the DCV 3DAA (Direct Acting Antiviral) Regimen) With or Without RBV for 12 Weeks for the Treatment of Chronic Hepatitis C Virus(HCV)Genotype 1 Infection in Subjects With Compensated Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AI443-113; 2013-002458-66 (EudraCT Number)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1: DCV/ASV/BMS-791325+Placebo matching RBV (naive) (Experimental): Triple fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg, BMS-791325 75 mg) tablet orally twice a day for 12 weeks
  Placebo matching Ribavirin 0mg tablet orally twice a day for 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir; Drug: BMS-791325; Drug: Placebo matching Ribavirin
- A2: DCV/ASV/BMS-791325 + RBV (naive) (Experimental): Triple fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg, BMS-791325 75 mg) tablet orally twice a day for 12 weeks
  Ribavirin 200mg tablet orally twice a day for 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir; Drug: BMS-791325; Drug: Ribavirin
- A3: DCV/ASV/BMS-791325+Placebo matching RBV (experienced) (Experimental): Triple fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg, BMS-791325 75 mg) tablet orally twice a day for 12 weeks
  Placebo matching Ribavirin 0 mg tablet orally twice a day for 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir; Drug: BMS-791325; Drug: Placebo matching Ribavirin
- A4: DCV/ASV/BMS-791325 + RBV (experienced) (Experimental): Triple fixed dose combination (Daclatasvir 30 mg, Asunaprevir 200 mg, BMS-791325 75 mg) tablet orally twice a day for 12 weeks
  Ribavirin 200 mg tablet orally twice a day for 12 weeks, Weight based dosing: If < 75 kg, 1000 mg per day (two 200 mg tablets in AM and three 200 mg tablets in PM); if ≥ 75 kg, 1200 mg per day (three 200 mg tablets in AM and three 200 mg tablets in PM), AM=in the morning, PM=in the evening
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir; Drug: BMS-791325; Drug: Ribavirin

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: BMS-790052
Drug: Asunaprevir
  Other Names: BMS-650032
Drug: BMS-791325
Drug: Ribavirin
  Other Names: Ribasphere®
  Arms: A2: DCV/ASV/BMS-791325 + RBV (naive); A4: DCV/ASV/BMS-791325 + RBV (experienced)
Drug: Placebo matching Ribavirin
  Arms: A1: DCV/ASV/BMS-791325+Placebo matching RBV (naive); A3: DCV/ASV/BMS-791325+Placebo matching RBV (experienced)

SUMMARY:
To demonstrate the effectiveness of DCV 3DAA fixed dose combination with or without Ribavirin in treatment naive cirrhotic subjects.

DETAILED DESCRIPTION:
Masking is Double blind for RBV: two or more parties are unaware of the intervention assignment.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects chronically infected with HCV genotype 1
* Subjects with compensated cirrhosis
* HCV RNA ≥ 10,000 IU/mL at screening
* Treatment-naïve subjects with no previous exposure to an interferon formulation (ie, IFNα, pegIFNα), Ribavirin (RBV), or HCV Direct Acting Antivirals (DAA) (protease, polymerase inhibitor, etc.)
* Treatment-experienced subjects are eligible including exposure to anti-HCV agents of a mechanistic class other than those contained in the Daclatasvir (DCV) / Asunaprevir (ASV) /BMS-791325 triple regimen is permitted. Examples of permitted agents include, but are not limited to nucleoside/nucleotide inhibitors of nonstructural protein 5B (NS5B) polymerase, inhibitors of cyclophilin, or inhibitors of microRNA.

Exclusion Criteria:

* Subjects without cirrhosis
* Liver or any other organ transplant
* Current or known history of cancer within 5 years prior to screening
* Documented or suspected hepatocellular carcinoma(HCC)
* Evidence of decompensated liver disease including, but not limited to, radiologic criteria, a history or presence of ascites, bleeding varices, or hepatic encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportion of treated subjects in each of the naive arms with sustained virologic response (SVR12) | Post treatment 12 week
  SVR12 is defined as Hepatitis C virus ribonucleic acid (HCV RNA) < Limit of Quantification (LOQ) target detected or target not detected (LOQ TD/TND)

SECONDARY OUTCOMES:
Proportion of treated subjects in each of the experienced arms with SVR12 | Post treatment 12 Week
Proportion of subjects in each arm who achieve HCV RNA < LOQ TD/TND | Weeks: 1, 2, 4, 6, 8, and 12; Post treatment Weeks 4 (SVR4), 8 (SVR8) and 24 (SVR24)
Proportion of subjects in each arm who achieve HCV RNA < LOQ TND | Weeks: 1, 2, 4, 6, 8, and 12; Post treatment Weeks 4 (SVR4), 8 (SVR8), 12 (SVR12) and 24 (SVR24)
Safety as measured by frequency of Serious Adverse Events(SAEs)and discontinuations due to Adverse Events(AEs) | Up to end of treatment (week 12) + 7 days
Proportion of subjects with anemia defined as Hg < 10 g/dL on-treatment and Hg ≥ 10 g/dL at baseline in each arm within each cohort | Up to end of treatment (week 12) + 7 days
Differences in rates of selected Grade 3 - 4 laboratory test result abnormalities | Up to end of treatment (week 12) + 7 days
Proportion of subjects achieving SVR12 associated with HCV geno subtype 1a vs 1b | Post treatment 12 Week
Proportion of subjects in each arm achieving SVR12 associated with IL28B rs12979860 single nucleotide polymorphism(SNP) status (CC genotype or non-CC genotype) | Post treatment 12 Week

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (44):
- United States (26):
  - Scripps Clinic, La Jolla, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University Of Colorado Denver & Hospital, Aurora, Colorado
  - Borland-Groover Clinic, Jacksonville, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Gastrointestinal Specialists Of Georgia, Marietta, Georgia
  - University Of Chicago, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Kansas City Care Clinic, Kansas City, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Binghamton Gastroenterology Associates, Binghamton, New York
  - Weill Cornell Medical College, New York, New York
  - Asheville Gastroenterology Associates, Pa, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Quality Medical Research Pllc, Nashville, Tennessee
  - Advanced Liver Therapies, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Mt Vernon Endoscopy Center, Alexandria, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Digestive And Liver Disease Specialists, Norfolk, Virginia
  - Dean Clinic, Madison, Wisconsin
- Australia (7):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Clayton, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Fremantle, Western Australia
- Canada (6):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Hamilton, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- France (5):
  - Local Institution, Créteil
  - Local Institution, Marseille
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Paris

REFERENCES:
- [Derived] Muir AJ, Poordad F, Lalezari J, Everson G, Dore GJ, Herring R, Sheikh A, Kwo P, Hezode C, Pockros PJ, Tran A, Yozviak J, Reau N, Ramji A, Stuart K, Thompson AJ, Vierling J, Freilich B, Cooper J, Ghesquiere W, Yang R, McPhee F, Hughes EA, Swenson ES, Yin PD. Daclatasvir in combination with asunaprevir and beclabuvir for hepatitis C virus genotype 1 infection with compensated cirrhosis. JAMA. 2015 May 5;313(17):1736-44. doi: 10.1001/jama.2015.3868. PMID 25942724
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx